CLINICAL TRIAL: NCT06420115
Title: AOP2780 - Can Needle Size Improve Cancer Detection Rate of Transperineal MRI Target Prostate Biopsy Without Affecting Side Effects?
Brief Title: Can Needle Size Improve Cancer Detection Rate of Transperineal MRI Target Prostate Biopsy Without Affecting Side Effects?
Acronym: TARGET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, FABIO ZATTONI, MD, Phd, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AOP2780
Record Dates: First submitted 2024-04-26; First posted 2024-05-17 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer Diagnosis
Keywords: pca; needle; 16 gauge; 18 gauge
MeSH Terms: conditions — Choanal Atresia, Posterior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mpMRI target prostate biopsy with 16 gauge needle (Experimental)
  Interventions: Device: different needle size for prostate biopsy
- mpMRI target prostate biopsy with 18 gauge needle (Experimental)
  Interventions: Device: different needle size for prostate biopsy

INTERVENTIONS:
Device: different needle size for prostate biopsy — MRI Fusion Transperineal Prostate Biopsy

SUMMARY:
Differences in terms of diagnostic capability and side effects related to the needle caliber used for prostate biopsy sampling in patients with suspected prostate cancer

DETAILED DESCRIPTION:
To assess whether a larger caliber (16G) prostate biopsy needle increases the diagnostic capability of prostate neoplasia compared to a smaller caliber (18G) needle, while keeping perioperative complications constant.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of prostate cancer (presence of elevated prostatic specific antigen and/or suspicious digital rectal examination);
* Presence of at least one suspicious prostate lesion on MRI (Prostate Imaging-Reporting and Data System ≥ 3) according to the Prostate Imaging-Reporting and Data System v2.1 performed before Magnetic Resonance Imaging/transrectal ultrasound fusion biopsy.

Exclusion Criteria:

* Patients under active surveillance or with a previous diagnosis of prostate neoplasia prior to biopsy.
* Previous radiotherapy to the prostate for neoplasia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Total number of random and fusion-target biopsies with presence of prostate cancer | When histological report available
  The primary outcome measure involves assessing the total number of biopsies, including both random and fusion-targeted approaches, that reveal the presence of prostate cancer.
Number of random and fusion-target biopsies with clinically significant prostate cancer (defined as International Society of Urological Pathology >=2) | When histological report available
  The primary outcome measure focuses on the number and the detection rates of random and fusion-target biopsies revealing clinically significant prostate cancer aof clinically significant prostate cancer (defined as ISUP >=2) between 16-gauge and 18-gauge biopsy needles.

SECONDARY OUTCOMES:
Neoplasia/core ratio for each random and fusion-target biopsy | When histological report available
  Neoplasia/core ratio, indicates the ratio of neoplastic tissue to healthy tissue within biopsy cores obtained through both 16 and 18 gauge biopsies for prostate cancer diagnosis. By analyzing this ratio, investivators seek to identify differences in diagnosis across the two different sizes
Intra- and perioperative pain with 18G and 16G needles assessed using visual analog scale (VAS) | 30 days
  The validated pain questionnaire employed in this study is designed to comprehensively assess the intra- and perioperative pain (following 7 days) experienced by patients undergoing prostate biopsy procedures with 18G and 16G needles. The visual analog scales "VAS" is a standardized validated questionnaire, a horizontal line, where one end represents "1 - no pain" and the other end represents "10 - worst possible pain." Patients are asked to mark on the line the point that best represents the intensity of their pain.
Number of hospitalizations at 30 and 60 days post-procedure | 60 days from biopsy
  By tracking the number of hospitalizations occurring at both 30 and 60 days post-procedure among patients undergoing prostate biopsy within these specific time frames, researchers seek to assess the short-term post-procedural outcomes and potential complications associated with the biopsy procedure. These hospitalization data will provide information into the safety profile and healthcare utilization patterns following prostate biopsy, aiding in the optimization of patient care and risk management strategies.
Number of intra- and perioperative complications associated with 18G and 16G needles | 30 days
  Intraoperative complications refer to adverse events occurring during the biopsy procedure itself, while perioperative complications encompass those arising in the immediate post-procedural period. These complications may include but are not limited to bleeding, infection, urinary retention, and vasovagal reactions. By documenting these complications, investigators will evaluate the safety profile and potential risks associated with each needle gauge, thereby informing clinical decision-making and optimizing patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Zattoni, MD, PhD, Principal Investigator — Department of Surgery, Oncology and Gastroenterology, Urology Clinic, University of Padua, Padova,
Locations (1):
- Urology Unit - Padua University Hospital, Padua, Italy, Italy

IPD SHARING:
Plan to Share IPD: No
Only if requested